CLINICAL TRIAL: NCT03276858
Title: A Double-Blind, Randomized, Placebo-Controlled, Single- And-Multiple-Dose Study to Evaluate the Safety, PK, and PD of CRN00808 in Healthy Volunteers and to Determine the Effect of CRN00808 on Midazolam PK
Brief Title: Single and Multiple-Ascending Dose Study of CRN00808 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRN00808-01
Record Dates: First submitted 2017-09-05; First posted 2017-09-08 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Single and multiple-dose cohorts are placebo-controlled. The midazolam cohort does not have placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CRN00808 Oral Solution (Experimental): CRN00808 oral solution, single-dose
  Interventions: Drug: CRN00808
- CRN00808 Oral Capsule (Experimental): CRN00808 oral capsule, single-dose and multiple-doses
  Interventions: Drug: CRN00808
- Placebo Oral Solution (Placebo Comparator): Placebo oral solution, single-dose
  Interventions: Drug: Placebo Oral Solution
- Placebo Oral Capsule (Placebo Comparator): Placebo oral capsule, single-dose and multiple doses
  Interventions: Drug: Placebo oral capsule
- Midazolam Oral Solution (Other): Midazolam oral solution, two single-doses as part of the drug-drug interaction arm of the study
  Interventions: Drug: CRN00808; Drug: Midazolam oral solution

INTERVENTIONS:
Drug: CRN00808 — Investigational drug
  Arms: CRN00808 Oral Capsule; CRN00808 Oral Solution; Midazolam Oral Solution
Drug: Placebo Oral Solution — Placebo
  Arms: Placebo Oral Solution
Drug: Midazolam oral solution — Midazolam as part of the drug-drug interaction arm of the study
  Arms: Midazolam Oral Solution
Drug: Placebo oral capsule — Placebo
  Arms: Placebo Oral Capsule

SUMMARY:
This single-center study will be conducted in 3 phases: a single-ascending dose phase (up to 8 cohorts, 8 subjects/cohort), a multiple-dose phase (up to 5 cohorts, 9 subjects/cohort), and a midazolam drug-drug interaction phase (one cohort of 8 subjects).

DETAILED DESCRIPTION:
The single-dose phase initiates with ascending doses of an oral solution followed by a 3-way crossover food effect and bioavailability (capsule formulation) cohort. Serum IGF-1 levels and GHRH-analog stimulated GH levels will be assessed as pharmacodynamics measures.

The first multiple-dose (7 days dosing) cohort will be initiated after the PK and safety data are available from the single-dose phase. Subsequent multiple-dose cohorts will have 10 days of dosing. Serum IGF-1 level and GH levels will be assessed as pharmacodynamics measures.

The last cohort in the study is midazolam drug-drug interaction study. The dose will be selected based on review of all pharmacokinetic and safety data for the single-dose and multiple-dose cohorts completed. On Day 1, 8 subjects will receive a single oral 2 mg dose of midazolam. Starting on Day 3 through Day 8, subjects will receive daily doses of CRN00808. On Day 9, subjects will be administered CRN00808 and 2 mg midazolam together.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18 to 30 kg/m2
* Females postmenopausal or surgically sterile

Exclusion Criteria:

* Any uncontrolled or active major systemic disease including, but not limited to: acromegaly (with or without pituitary surgery or radiation therapy), cardiac, pulmonary, gastrointestinal, metabolic, urogenital, neurological, immunological, psychiatric, or neoplastic disorder with metastatic potential
* History or presence of malignancy within the past 5 years. Subjects who have been successfully treated (for 3 months or longer) with no recurrence of basal or squamous cell carcinoma of the skin or carcinoma in-situ of the cervix may be enrolled.
* Use of any investigational drug within the past 60 days or 5 half-lives, whichever is longer
* Have a medically significant abnormality observed during screening or the admission physical examination or in any other baseline measurements
* Use of any prior medication without approval of the investigator within 14 days prior to admission
* Tested positive at screening for HIV, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV-Ab) or has a history of a positive result
* History of alcohol or substance abuse in the past 6 months
* Any condition that in the opinion of the investigator would jeopardize the subject's appropriate participation in this Phase 1 study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of CRN00808 single ascending doses using clinical assessments, telemetry, and Holter monitoring and subject self-reporting | Day 1 through Day 10
  ECG, clinical laboratory parameters, vital signs, physical examinations, telemetry, Holter monitoring
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of CRN00808 multiple ascending doses using clinical assessments and subject self-reporting | Day 1 through Day 21
  ECG, clinical laboratory parameters, vital signs, physical examinations

SECONDARY OUTCOMES:
AUC of CRN00808 single ascending doses | Day 1 through Day 7
  plasma AUC
Cmax of CRN00808 single ascending doses | Day 1 through Day 7
  plasma Cmax
t1/2 of CRN00808 single ascending doses | Day 1 through Day 7
  plasma t1/2
Tmax of CRN00808 single ascending doses | Day 1 through Day 7
  plasma Tmax
AUC of CRN00808 multiple ascending doses | Day 1 through Day 20
  plasma AUC
Cmax of CRN00808 multiple ascending doses | Day 1 through Day 20
  plasma Cmax
t1/2 of CRN00808 multiple ascending doses | Day 1 through Day 20
  plasma t1/2
Tmax of CRN00808 multiple ascending doses | Day 1 through Day 20
  plasma Tmax
Pharmacodynamics of CRN00808 in single ascending dose cohorts assessed by GHRH analog stimulated GH levels | Day -1 and Day 1
  Suppression of serum GH induced by a GH secretagogue
Effect of CRN00808 on pharmacokinetics of midazolam | Day 1 through Day 10
  midazolam plasma AUC
Effect of CRN00808 on Cmax of midazolam | Day 1 through Day 10
  midazolam plasma Cmax
Effect of CRN00808 on t1/2 of midazolam | Day 1 through Day 10
  midazolam plasma t 1/2
Effect of CRN00808 on Tmax of midazolam | Day 1 through Day 10
  midazolam plasma Tmax
Relative bioavailability of capsule formulation | Day 1 to Day 7
  single-dose crossover arm only
Effect of food on Cmax of CRN00808 | Day 1 to Day 7
  plasma Cmax compared with and without food in single dose arm
Effect of food on AUC of CRN00808 | Day 1 to Day 7
  Plasma AUC compared with and without food in single dose arm
Pharmacodynamics of CRN00808 in multiple ascending dose cohorts assessed by serum IGF-1 and GH | Day -1 to Day 21
  serum IGF-1 and GH

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MBBS PhD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madan A, Markison S, Betz SF, Krasner A, Luo R, Jochelson T, Lickliter J, Struthers RS. Paltusotine, a novel oral once-daily nonpeptide SST2 receptor agonist, suppresses GH and IGF-1 in healthy volunteers. Pituitary. 2022 Apr;25(2):328-339. doi: 10.1007/s11102-021-01201-z. Epub 2022 Jan 9. PMID 35000098